CLINICAL TRIAL: NCT05821634
Title: Digital Phenotyping of Anxiety and Anxiety-Related Alcohol Comorbidity and Treatment
Brief Title: Personalizing Treatment Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Marilyn L. Piccirillo, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00013899; 4R00AA029459-03 (NIH)
Record Dates: First submitted 2023-03-26; First posted 2023-04-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Anxiety Disorders and Symptoms; PTSD and Trauma-related Symptoms; Alcohol; Use, Problem; Alcohol Use Disorder
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized intervention condition (Experimental): This experimental condition will test a data-driven, person-specific intervention using CBT skills.
  Interventions: Behavioral: Personalized intervention condition: Cognitive behavioral therapy skills
- Therapeutic control condition (Active Comparator): This control condition will provide an experimental comparison to test the process of personalization.
  Interventions: Behavioral: Therapeutic control condition: Cognitive behavioral therapy skills
- Tracking control condition (Active Comparator): This second control condition will provide an experimental comparison to test the effects of health-related tracking and therapeutic contact.
  Interventions: Behavioral: Tracking control condition: Supportive counseling

INTERVENTIONS:
Behavioral: Personalized intervention condition: Cognitive behavioral therapy skills — An 11-session cognitive behavioral therapy (CBT) skills based intervention will be delivered to participants randomized to the personalized intervention. Influential constructs will be identified using the person specific digital phenotyping model, targeted using CBT skills, and tracked across sessions.
  Arms: Personalized intervention condition
Behavioral: Therapeutic control condition: Cognitive behavioral therapy skills — Participants randomized to this condition will receive an 11-session CBT skills based treatment targeting a non-personalized construct selected from the person-specific digital phenotyping model.
  Arms: Therapeutic control condition
Behavioral: Tracking control condition: Supportive counseling — Participants randomized to this condition will receive 11 supportive counseling sessions that are non-directive in nature (providing support and validation for non-acute weekly stressors). Participants will continue digital phenotyping, controlling for the effect of counseling and digital phenotyping.
  Arms: Tracking control condition

SUMMARY:
Anxiety and anxiety-related disorders frequently co-occur with alcohol use problems resulting in an enormous humanitarian and economic cost to society. The proposed research will use digital technology to examine person-specific risk factors predicting problematic alcohol use in individuals vulnerable to anxiety and anxiety-related disorders and will use this information to design a personalized intervention for individuals seeking psychological treatment. Results from this research will integrate output from novel and innovative digital technology methods into psychotherapy, advancing research on personalized treatment and prevention efforts.

ELIGIBILITY:
Inclusion Criteria:

* Access to a smart phone
* Between 18 and 65 years
* Clinically significant anxiety or trauma-related symptoms
* Alcohol use problems
* Interest in telehealth counseling
* Anticipated New Jersey or New York residence for the duration of the study

Exclusion Criteria:

* Currently receiving counseling
* Psychiatric medication that is not currently at a stable dose (or is not anticipated to remain at a stable dose for the duration of the study)
* Demonstrated indicators of more intensive or acute care
* Temporary residence within the state of New Jersey or New York or out-of-state residence from the state of New Jersey or New York

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol related risk | Week 3, Week 15 (approximate)
  The Alcohol Use Disorder Identification Test (AUDIT) self-report measure (or similar) will be used to assess changes in alcohol related risk.
Change in risk drinking levels | Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Week 13, Week 14, Week 15 (approximate)
  The Daily Drinking Questionnaire (DDQ) self-report measure (or similar) will be used to measure changes in alcohol consumption/risk drinking levels.
Change in anxiety or anxiety-related symptom severity | Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Week 13, Week 14, Week 15 (approximate)
  The Overall Anxiety Severity and Impairment Scale (OASIS) self-report measure (or similar) will be used to assess changes in anxiety and anxiety-related symptom severity.
Change in psychiatric diagnoses | Week 3, Week 15 (approximate)
  A diagnostic interview will be used to assess change in psychiatric diagnoses at the beginning and end of participation.

SECONDARY OUTCOMES:
Number of sessions attended | Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Week 13, Week 14, Week 15 (approximate)
  The number of sessions completed (up to 11) will be used to measure treatment engagement.
Change in therapeutic alliance | Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Week 13, Week 14, Week 15 (approximate)
  The Working Alliance Inventory self-report measure (or similar) will be used to measure changes in working therapeutic alliance.
Patient-rated assessment of progress | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Week 13, Week 14, Week 15 (approximate)
  Patient-rated improvements in functioning assessed will be assessed at (approximately) weekly intervals.
Clinician-rated improvement in functioning | Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, Week 13, Week 14, Week 15 (approximate)
  Clinician-rated improvements in functioning assessed will be assessed at the beginning and end of study participation, as well as at (approximately) weekly intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Piccirillo, PhD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided